CLINICAL TRIAL: NCT06483607
Title: Comparison of the Analgesic Effects of Modified Thoracoabdominal Nerve Block Through Pericondrial Approach (M-TAPA) and Transversus Abdominis Plane (TAP) Block in Laparoscopic Inguinal Hernia Surgeries
Brief Title: Comparison of M-TAPA and TAP Blocks on Postoperative Analgesia in Laparoscopic Inguinal Hernia Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Associate Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Comparison of M-TAPA and TAP
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Post Operative Pain
Keywords: m-tapa; tap block; laparoscopic inguinal hernia; regional anesthesia; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL (No Intervention): Control group patients are not going to be subjected to any block or local infiltration anesthesia. Their postoperative pain will be relieved with ibuprofen and tramadol (intravenous) administrations.
- M-TAPA (Active Comparator): Patients will have bilateral M-TAPA block with 0.25% bupivacaine (total volume of 40 ml) at the end of the surgery for postoperative pain control.
  Interventions: Other: M-TAPA block with bupivacaine 25%
- TAP (Active Comparator): Patients will have bilateral lateral-TAP block with 0.25% bupivacaine (total volume of 40 ml) at the end of the surgery for postoperative pain control.
  Interventions: Other: TAP block with bupivacaine 25%

INTERVENTIONS:
Other: M-TAPA block with bupivacaine 25% — Following sterile conditions for bilateral M-TAPA block application, the transducer will be inserted on the chondrium in the sagittal plane at the 9-10th rib level. Subsequently, a deep angle will be created with the probe for visualization of the underside of the costochondrium. The sonovisible needle tip will be placed just below the chondrium and saline (5 ml) will be injected for site confirmation. After the confirmation, 20 ml of 0.25% bupivacaine will be administered for each group for a total of 40 ml of local anesthetic. Blocks will be applied using an 80 mm sonovisible needle with a 6-10 MHz linear probe under the guidance of a portable ultrasound. M-TAPA block with the same standard technique and drug dose will be applied to the contralateral side for each group of M-TAPA patients.
  Other Names: Modified thoracoabdominal nerve block through perichondrial approach
  Arms: M-TAPA
Other: TAP block with bupivacaine 25% — After the necessary sterilization conditions established, the linear ultrasound probe will be placed in the middle of the iliac crest with the end limit of the ribs. Starting with skin, the layers in descending order, subcutaneous adipose tissue, external oblique muscle, internal oblique muscle, transversus abdominis muscle, and peritoneum will be identified. As the tip of the 80 mm sonovisible needle passes through the muscular layers and fascia, the needle will be advanced in a controlled manner. After receiving the click sensation (passage of the fascia of the internal oblique muscle), the location of the needle will be fixed and 20 ml of 0.25% bupivacaine will be injected between internal oblique and transversus abdominis muscles. Same procedure will be performed to the other site. (40 ml local anesthetics in total)
  Other Names: Transversus abdominis plane block
  Arms: TAP

SUMMARY:
The goal of this study is to compare the analgesic efficacy of M-TAPA block and TAP block in patients undergoing laparoscopic inguinal hernia surgeries.

DETAILED DESCRIPTION:
There will be three randomized groups: Group Control (no any block, n=30) Group M-TAPA (n=30), Group TAP (n=30). All patients will have standard general anesthesia. Group M-TAPA patients will receive bilateral M-TAPA block with 0.25% bupivacaine (total volume of 40 ml). Group TAP patients will have bilateral lateral-TAP block with 0.25% bupivacaine (total volume of 40 ml). All blocks will be performed at the end of the surgery, before awakening the patients. All patients in the study will receive 50 mg dexketoprofen and 1 gr paracetamol intravenos (i.v.) 10 minutes prior to skin closure. All patients will have ibuprofen 3x400 mg in postoperative 24 hours (maximum dose 1200 mg/day). Numerical rating scale (NRS) will be used to assess postoperative pain on 1st, 6th, 12th, 18th and 24th hour after the surgery. 50 mg tramadol will be administered as a rescue analgesic in all patients.Total tramadol consumption will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 18 years of age who will undergo laparoscopic inguinal hernia under general anesthesia and will be American Society of Anesthesiologists (ASA) I-II-III according to the ASA risk classification.

Exclusion Criteria:

* Patients who did not give consent,
* patients with coagulopathy,
* patients with signs of infection at the block application site,
* patients using anticoagulants,
* patients with local anesthetic drug allergies,
* patients undergoing open surgery,
* patients with unstable hemodynamics,
* patients who could not cooperate during postoperative pain assessment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2026-01-17 (Actual)

PRIMARY OUTCOMES:
Comparing the numerical rating scale scores | Postoperative 24 hours
  Numerical rating scale will be used for pain assessment. The scores of the numerical rating scale changes between 0 to 10 points. 10 points mean "the most severe pain that the patient ever had". 0 point means "there is no pain." Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Comparing total tramadol consumption | Postoperative 24 hours
  Postoperative analgesic need

CONTACTS AND LOCATIONS:
Overall Officials: Oğuz Gündoğdu, Principal Investigator — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation
Locations (1):
- Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation, Sivas, Si̇vas, Turkey (Türkiye)